CLINICAL TRIAL: NCT06380634
Title: Gebelikte Ev İçi Kimyasallar ve Kişisel Bakım Ürünlerinin Kullanımını Azaltmada Motivasyonel Görüşmenin Etkinliği
Brief Title: The Effectiveness of Motivational Interviewing in Reducing the Use of Household Chemicals and Personal Care Products During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Nazli Yalcinbas, midwife, Istanbul University - Cerrahpasa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: NYalcinbas
Record Dates: First submitted 2024-03-12; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Motivational Interview; Cosmetic Product Causing Toxic Effect
Keywords: Household Product; Midwifery; Pregnancy

STUDY DESIGN:
Intervention Model Description: The research was conducted in a prospective pre-test, post-test based randomized controlled experimental research design.
Masking Description: The groups were randomized into 2 groups using a web-based randomization program (http://www.randomizer.org). The researcher included pregnant women who met the inclusion criteria in the outpatient clinics on certain days of the week, in accordance with the randomization process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Randomize) (Experimental): The sample size was determined as at least 64 people for each of the experimental and control groups, with 80% power, 0.05 margin of error and 0.5 effect level. Considering the possibility of data loss later on, 70 pregnant women (140 in total) were included in each group. The groups were randomized into 2 groups using a web-based randomization program (http://www.randomizer.org). 357 pregnant women were evaluated for suitability for the study. 68 women did not meet the inclusion criteria and 149 women were not included because they did not agree to participate in the study. The pre-test of the study was completed with 70 experimental and 70 control groups (140 in total), and the post-test was completed with a total of 130 people, 69 experimental and 61 control groups.
  Interventions: Behavioral: Experimental group- Motivational Interview

INTERVENTIONS:
Behavioral: Experimental group- Motivational Interview — Pregnant women who applied to the gynecology clinic and met the inclusion criteria were informed about the study. Those who agreed were informed about the purpose of the research. Firstly, the Informed Volunteer and Introductory Information Form was applied to the women, then the Personal Care Products Use Evaluation Form, Self-Efficacy Scale and Endocrine Disruptors Attitude Scale were applied. Then, the experimental group was informed about the motivational interviewing technique. A total of 3 interviews were held. The final test was made at the fourth meeting.

SUMMARY:
Objective: The aim of the study is to examine the effect of motivational interviewing on reducing the use of household chemicals and personal care products during pregnancy.

DETAILED DESCRIPTION:
Introduction :During pregnancy, women are exposed to cosmetic products and household chemicals frequently used in daily life.

Method: The research was conducted in a prospective pre-test, post-test based randomized controlled experimental research design.The sample of the study consisted of 140 pregnant women who applied to the Ministry of Health Istanbul Provincial Health Directorate and Sile State Hospital Gynecology and Obstetrics Polyclinics between May and December 2023, volunteered to participate in the study and met the inclusion criteria.

Firstly, the Informed Consent Form and Introductory Information Form were applied to the women, then the Personal Care Products Use Evaluation Form, Self-Efficacy Scale and Endocrine Disruptors Attitude Scale were applied. The experimental group was informed about the motivational interviewing technique and an appropriate plan was made. After the interviews, the Personal Care Products Use Evaluation Form, Self-Efficacy Scale and Endocrine Disruptors Attitude Scale were re-administered.

ELIGIBILITY:
Inclusion Criteria:

* Being at least 18 years old
* Education level must be at least primary school
* Speaking Turkish
* Having a single pregnancy between the 8th and 40th weeks
* Using household chemicals and personal care products (any product at least once a week)

Exclusion Criteria:

* Having a psychiatric illness that prevents communication,
* Having a chronic serious physical health problem
* Termination of pregnancy for any reason
* Having a risky pregnancy (preeclampsia, threat of premature birth)
* Intrauterine growth retardation, having a pregnancy with fetal anomalies
* Working in a job that requires heavy use of chemicals, such as hairdresser, dry cleaner, beautician.

Ages: 20 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 130 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Evaluation Form for Use of Domestic Chemicals and Personal Care Products | 1 year
  In this form prepared by the researcher in line with the literature, the use of cosmetic products was asked with 41 product names in five main categories such as rinsed products, products applied to the skin and not rinsed, products applied to the hair, make-up products, intimate care products; Household chemicals are asked with 12 product names (Ashrap et al., 2018; Ingle et al., 2019; Preston et al., 2021; Fruh et al., 2022; Deierlein et al., 2022). The personal care product usage frequency of the experimental and control groups was asked in a 5-point Likert type at the pre-test and post-test, and then the difference in pre-test and post-test product usage was categorized as increasing, remaining the same or decreasing.
Self Efficacy Competence Scale | 1 year
  On a five-point Likert-type scale consisting of 23 items, each item is marked as 1-does not describe me at all, 2-describes me a little, 3-undecided, 4-describes me well, 5-describes me very well.
Endocrine Disruptors Attitude Scale | 1 year
  The scale consists of 21 items. The endocrine disruptors attitude scale has two sub-dimensions: consumer behavior and nutrition and hygiene. The scale was prepared as a five-point Likert type as "I completely agree", "I agree", "I am undecided", "I disagree", "I strongly disagree".

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Preston EV, Chan M, Nozhenko K, Bellavia A, Grenon MC, Cantonwine DE, McElrath TF, James-Todd T. Socioeconomic and racial/ethnic differences in use of endocrine-disrupting chemical-associated personal care product categories among pregnant women. Environ Res. 2021 Jul;198:111212. doi: 10.1016/j.envres.2021.111212. Epub 2021 May 3. PMID 33957140
- [Background] Deierlein AL, Grayon AR, Zhu X, Sun Y, Liu X, Kohlasch K, Stein CR. Personal Care and Household Cleaning Product Use among Pregnant Women and New Mothers during the COVID-19 Pandemic. Int J Environ Res Public Health. 2022 May 6;19(9):5645. doi: 10.3390/ijerph19095645. PMID 35565038
- [Background] Ashrap P, Watkins DJ, Calafat AM, Ye X, Rosario Z, Brown P, Velez-Vega CM, Alshawabkeh A, Cordero JF, Meeker JD. Elevated concentrations of urinary triclocarban, phenol and paraben among pregnant women in Northern Puerto Rico: Predictors and trends. Environ Int. 2018 Dec;121(Pt 1):990-1002. doi: 10.1016/j.envint.2018.08.020. Epub 2018 Oct 11. PMID 30316544
- [Background] Fruh V, Preston EV, Quinn MR, Hacker MR, Wylie BJ, O'Brien K, Hauser R, James-Todd T, Mahalingaiah S. Urinary phthalate metabolite concentrations and personal care product use during pregnancy - Results of a pilot study. Sci Total Environ. 2022 Aug 20;835:155439. doi: 10.1016/j.scitotenv.2022.155439. Epub 2022 Apr 22. PMID 35469886
- [Background] Ingle ME, Watkins D, Rosario Z, Velez Vega CM, Huerta-Montanez G, Calafat AM, Ospina M, Cordero JF, Alshawabkeh A, Meeker JD. The association of urinary organophosphate ester metabolites and self-reported personal care and household product use among pregnant women in Puerto Rico. Environ Res. 2019 Dec;179(Pt A):108756. doi: 10.1016/j.envres.2019.108756. Epub 2019 Sep 23. PMID 31574449

DOCUMENTS (3):
  • Study Protocol (2024-02-05): https://cdn.clinicaltrials.gov/large-docs/34/NCT06380634/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-05): https://cdn.clinicaltrials.gov/large-docs/34/NCT06380634/SAP_001.pdf
  • Informed Consent Form (2023-12-30): https://cdn.clinicaltrials.gov/large-docs/34/NCT06380634/ICF_002.pdf